CLINICAL TRIAL: NCT05616793
Title: An Open Label, Dose Exploration, Safety and Tolerability Study of a Subretinal Injection of an OPGx-001 Gene Vector to Participants With LCA5-Associated Inherited Retinal Degeneration (LCA5-IRD) With OCncurrent Non-Interventional Follow-Up of Untreated Patients
Brief Title: Safety and Tolerability Subretinal OPGx-001 for LCA5-Associated Inherited Retinal Degeneration (LCA5-IRD) and Non-interventional Arm With Untreated Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Opus Genetics, Inc (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPGx-LCA5-1001; FD-R-008174 (Other Grant/Funding Number: Funding Source- FDA Office of Orphan Product Development (OOPD) Grant)
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: LCA5
Keywords: LCA; Retinal Degeneration; IRD; adeno associated virus; gene therapy; LCA5
MeSH Terms: conditions — Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: Enrollment will begin with a low-dose of OPGx-001 delivered via single, unilateral subretinal injection (Cohort 1) and proceed to an intermediate dose (Cohort 2) and subsequent high dose (Cohort 3). Escalation to each next cohort will proceed only after review of all data and upon recommendation by an independent data monitoring committee (IDMC).
  Concurrently, 16 untreated patients will be assessed for 6 months prior to treatment to study the natural course of LCA5-IRD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Group 1 (Experimental): A single, unilateral, subretinal injection of low dose (1E10 vg/eye) OPGx-001 is injected into two LCA5 adults (18 yo or above) in a sentinel fashion. A 30-day safety evaluation and data committee review and approval of continued dosing occurs. If additional dosing is recommended, a subsequent LCA5 adolescent (13-17) may be treated in a sentinel fashion, with a unilateral, subretinal injection of OPGx-001. A 30-day safety evaluation and data committee review and approval of continued dosing occurs. If additional dosing is recommended, two remaining adolescents (13-17) are eligible to be treated with a single, unilateral, subretinal injection of a low dose of OPGx-001. Total cohort size is 5 (2 adults and 3 adolescents).
  Interventions: Biological: AAV8.hLCA5
- Dose Group 2 (Experimental): A single, unilateral, subretinal injection of an intermediate dose (3E10 vg/eye) OPGx-001 is injected into two LCA5 adults (18 yo or above) in a sentinel fashion. A 30-day safety evaluation and data committee review and approval of continued dosing occurs. If additional dosing is recommended, a subsequent LCA5 adolescent (13-17) may be treated in a sentinel fashion, with a unilateral, subretinal injection of OPGx-001. A 30-day safety evaluation and data committee review and approval of continued dosing occurs. If additional dosing is recommended, two remaining adolescents (13-17) are eligible to be treated with a single, unilateral, subretinal injection of an intermediate dose of OPGx-001. Total cohort size is 5 (2 adults and 3 adolescents).
  Interventions: Biological: AAV8.hLCA5
- Dose Group 3 (Experimental): A single, unilateral, subretinal injection of high dose (1E11 vg/eye) OPGx-001 is injected into two LCA5 adults (18 yo or above) in a sentinel fashion. A 30-day safety evaluation and data committee review and approval of continued dosing occurs. If additional dosing is recommended, a subsequent LCA5 adolescent (13-17) may be treated in a sentinel fashion, with a unilateral, subretinal injection of OPGx-001. A 30-day safety evaluation and data committee review and approval of continued dosing occurs. If additional dosing is recommended, two remaining adolescents (13-17) are eligible to be treated with a single, unilateral, subretinal injection of a high dose of OPGx-001. Total cohort size is 5 (2 adults and 3 adolescents).
  Interventions: Biological: AAV8.hLCA5
- Part B Observational (No Intervention): Part B will occur concurrently with Dose Groups 1-3. Sixteen patients will be assessed for 6 months to assess the natural course of LCA5-IRD, then will be treated with OPGx-001 which will be described in a future protocol amendment.

INTERVENTIONS:
Biological: AAV8.hLCA5 — Adeno-associated virus vector expressing human LCA5 gene
  Arms: Dose Group 1; Dose Group 2; Dose Group 3

SUMMARY:
The goals of this clinical trial are assess the natural course of LCA5-IRD over 6 months and to evaluate the safety and preliminary efficacy of subretinal gene therapy with OPGx-001 in patients with inherited retinal degeneration due to biallelic mutations in the LCA5 gene. Funding Source- FDA Office of Orphan Products Development (OOPD).

DETAILED DESCRIPTION:
This is a non-randomized, open-label, phase 1/2 dose-escalation study evaluating untreated patients for 6 months and with three doses of OPGx-001 for the treatment of LCA5-IRD.

Enrollment will begin with a low-dose of OPGx-001 delivered via single, unilateral subretinal injection (Cohort 1) and proceed to an intermediate dose (Cohort 2) and subsequent high dose (Cohort 3). Escalation to each next cohort will proceed only after review of all data and upon recommendation by an independent data monitoring committee (IDMC).

Concurrently, 16 untreated patients will be assessed for 6 months prior to treatment to study the natural course of LCA5-IRD.

ELIGIBILITY:
Inclusion Criteria:

1. Are willing and able to provide written informed consent (ICF) and, where appropriate, willing to sign an assent prior to any study procedures.
2. Are willing to adhere to the clinical protocol and able to perform testing procedures.
3. In part A participants must be 13 years of age or older at consent, for Part B, participants must be 4 years of age or older at consent with the ability to conduct the MLoMT.
4. Carry disease-causing biallelic LCA5 gene mutations determined by a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory (historic testing up to 15 years from date of consent can be considered).
5. Visual acuity: BCVA < 20/80 on the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity chart (modified for low vision participants) in the eye to be treated
6. Show evidence of detectable photoreceptors by Spectral Domain Optical Coherence Tomography (SD-OCT)
7. Participant is a good candidate for surgery per investigator judgement
8. Participant agrees to follow direction of investigator regarding restrictions post-surgery (Part A only).

Exclusion Criteria:

1. Women who are pregnant or individuals (women of childbearing potential and men) unwilling to use effective contraception for the duration of the study, including barrier methods for the first year after investigational product (IP) administration (Part A only).
2. Pre-existing eye conditions or complicating systemic diseases that would preclude the planned surgery. This includes individuals who are immunocompromised.
3. History of intraocular surgery for either eye within 6 months prior to planned IP administration (Part A only).
4. Have previously received gene therapy.
5. Have used any investigational drug or device within 90 days or 5 estimated half-lives of treatment, whichever is longer or plan to participate in another study of drug or device during the study period.
6. History of disease which may preclude the participant from participation, or which may interfere with outcome measure testing or test results.
7. Incapable of performing visual function testing (e.g., FST testing) for reasons other than poor vision.
8. Any absolute contraindication to a course of oral steroids.
9. Any other condition that would not allow the potential participant to complete follow-up examinations during the study and, in the opinion of the Investigator, makes the potential participant unsuitable for the study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | 2 years
  Number of DLT events
Number of adverse events related to OPGx-001 | 2 years
  Number of AEs related to IP
Incidence of adverse events related to OPGx-001 | 2 years
  Incidence of AEs related to IP
Severity of adverse events related to OPGx-001 | 2 years
  Severity of AEs related to IP
Number of procedure-related adverse events | 2 years
  Number of AEs related to IP administration
Incidence of procedure-related adverse events | 2 years
  Incidence of AEs related to IP administration
Severity of procedure-related adverse events | 2 years
  Severity of AEs related to IP administration
Assessment of cross-sectional spectral domain optical coherence tomography images | 2 years
  Qualitative Assessment of SD-OCT image
Assessment of Natural course of LCA5-IRD | 6 months
  Change from baseline in MLoMT
Assessment of Natural course of LCA5-IRD | 6 months
  Change from baseline in FST
Assessment of Natural course of LCA5-IRD | 6 months
  Change from baseline in BCVA
Assessment of Natural course of LCA5-IRD | 6 months
  Change from baseline in FCP/Microperimetry
Assessment of Natural course of LCA5-IRD | 6 months
  Change from baseline in SD-OCT
Assessment of Natural course of LCA5-IRD | 6 months
  Change from baseline in pupillometry
Assessment of Natural course of LCA5-IRD | 6 months
  Number of adverse events

SECONDARY OUTCOMES:
Change from baseline over time in Multi-luminance Orientation and Mobility Test | 2 years
  Number of objects identified
Change from baseline over time in Dark-adapted full-field sensitivity testing | 2 years
  FST
Change from baseline over time in best corrected visual acuity (BCVA) | 2 years
  Measured using LogMAR scale
Change from baseline over time in visual functioning questionnaire | 1 year
  Assessed by the Modified National Eye Institute Visual Functioning Questionnaire

OTHER OUTCOMES:
Microperimetry | 1 year
  Mean sensitivity, in dB
Kinetic perimetry | 1 year
  Field extent, in degrees
Virtual Reality Orientation and Mobility Test (VR-O&M) | 1 year
  Performance over a range of light levels
Frequency doubling technology (FDT) perimetry (sFDT-CA) | 1 year
Light-adapted transient pupillary light reflex (LA-TPLR) | 1 year
Sweep visual evoked potentials (sVEPs) | 1 year
Chromatic referential looking | 1 year
  In dark-adapted patients
Full-field chromatic sensitivity testing (FST) | 1 year
  In free view
Portable chromatic pupillometry Portable chromatic pupillometry | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Retina Foundation of the Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No